CLINICAL TRIAL: NCT01361399
Title: A 4-arm, Multicenter, Randomized, Double-blind, Placebo- and Active-controlled, Single Dose, Parallel Group Study Comparing Efficacy and Safety of a Fixed Combination of 500 mg Acetylsalicylic Acid + 4 mg Lidocaine With 500 mg Acetylsalicylic Acid and 4 mg Lidocaine Monotherapy as Well as Placebo in Adult Patients With Sore Throat Associated With a Common Cold.
Brief Title: Active and Placebo Controlled Study to Test the Efficacy and Safety of an Aspirin-Lidocaine Lozenge in the Symptomatic Treatment of Sore Throat Associated With a Common Cold
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11640
Record Dates: First submitted 2011-05-25; First posted 2011-05-26 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Common Cold; Pharyngitis; Tonsillitis
Keywords: Sore Throat
MeSH Terms: conditions — Common Cold; Pharyngitis; Tonsillitis | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Acetylsalicylic acid (Aspirin, BAYE4465) & Lidocain
- Arm 2 (Active Comparator)
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)
- Arm 3 (Active Comparator)
  Interventions: Drug: Lidocain
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic acid (Aspirin, BAYE4465) & Lidocain — Single oral application of a fixed combination of Aspirin and Lidocain (as one lozenge)
  Arms: Arm 1
Drug: Acetylsalicylic Acid (Aspirin, BAYE4465) — Single oral application of Aspirin (as lozenge)
  Arms: Arm 2
Drug: Lidocain — Single oral application of Lidocain (as lozenge)
  Arms: Arm 3
Drug: Placebo — Single oral application of Placebo (as lozenge)
  Arms: Arm 4

SUMMARY:
The purpose of this study is to investigate the analgesic efficacy of a single dose of a fixed combination of 500 mg Aspirin (Acetylsalicylic Acid) and 4 mg Lidocaine in adult patients with sore throat associated with a common cold in comparison to a single treatment with 500 mg Aspirin or 4 mg Lidocaine alone as well a Placebo (treatment without any active ingredient). The combination of Aspirin and Lidocaine in a single lozenge is expected to provide relief from sore throat pain by sequential action. A very fast inset of action will be achieved by the locally acting Lidocaine and a long duration of action will be achieved by the systemically acting Aspirin.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of at least 18 years of age
* Onset of common cold within the last 3 days (12 to 72 hours)
* History of at least 4 symptoms associated with URTI in the last 24 hours out of runny nose, stuffy nose, sneezing, wet cough, dry cough, sweating, earache, ear fullness, sinus pressure/pain, head heaviness, muscle aches and pains, feverish discomfort, chills, hoarseness, sore throat, scratchy throat and headache as documented in the history of URTI
* Current sore throat confirmed by a score ≥ 6 on a 11-category vertical ordinal scale for sore throat pain
* Findings that confirmed the presence of tonsillopharyngitis

Exclusion Criteria:

* Pregnancy (i.e. positive pregnancy test at baseline)
* Breastfeeding
* History of hypersensitivity (allergic reaction) to ASA or any other NSAID
* History of hypersensitivity (allergic reaction) to lidocaine
* History or acute state of peptic ulceration or gastrointestinal bleeding
* History of bleeding tendency
* History of asthma
* Clinical diagnosis of chickenpox or influenza
* History or presence of severe liver or kidney disease
* Intake of short-acting analgesics (e.g. ASA, paracetamol, ibuprofen, diclofenac) either as a single ingredient or as part of a combination cold product in the last 6 hours, or intake of long-acting analgesics (e.g. naproxen) in the last 12 hours, or intake of any other NSAID in the last 24 hours
* Use of any local or systemic short-acting cough and cold preparation (e.g. decongestant or antihistaminic drug) in the last 12 hours
* Use of any cough or sore throat lozenges/candies or any menthol-containing product (including mentholated tissues) in the last 6 hours
* Current intake or requirement of any prescription medication for the current treatment of acute respiratory tract illness
* Administration of anticoagulants in the last 7 days
* Inability to breathe through the nose or a history of chronic mouth breathing
* Presence of any severe concomitant disease or condition which, in the opinion of the investigator, is a reason for exclusion, e.g. serious cardiovascular diseases (in particular arrhythmias), treatment with antiarrhythmics or methotrexate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1088 (Actual)
Dates: Start 2004-11-30 (Actual); Primary Completion 2005-05-28 (Actual); Study Completion 2005-05-28 (Actual)

PRIMARY OUTCOMES:
Sum of pain intensity differences SPID | 120 minutes
Pain intensity difference to baseline (PID12 min) | 12 minutes
Pain intensity difference to baseline (PID120 min) | 120 minutes

SECONDARY OUTCOMES:
Pain intensity difference to baseline (PID) | 3, 6, 12, 18, 24, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 and 240 minutes post dose
Total pain relief to baseline (TOTPAR) | 3, 6, 12, 18, 24, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 and 240 minutes post dose
Symptoms of common cold (headache, sinus pressure/pain, feverish discomfort, muscle aches and pain) | 60, 120, 180, and 240 minutes post dose
Overall assessment of treatment | 240 minutes
Assessment of safety and tolerability | 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer; Bayer Study Director — Bayer
Locations (5):
- Russia (3):
  - Mocow
  - Moscow
  - Novosibirsk
- Ukraine (2):
  - Kiev
  - Luhansk